CLINICAL TRIAL: NCT05404269
Title: Comparison of AGC (Automatic Gas Control) Mode and Manually Controlled Minimal Flow Anesthesia in Breast Surgery
Brief Title: AGC Mode vs Minimal Flow in Breast Surgery
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Gökhan Çeviker, Anesthesiologist, Zonguldak Bulent Ecevit University
Other Study IDs: 2021/05-12
Record Dates: First submitted 2022-05-30; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Volatil Agent Consumption; Automatic End-tidal Controlled Anesthesia; Anesthesia; Functional; Breast Diseases
Keywords: anesthesia machine; sevoflurane; minimal fresh gas flow; breast surgery; AGC mode
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group AGC: The FLOW-i anesthesia machine (Maquet, Solna, Sweden) can be equipped with automated gas control (AGC), an automated low flow tool with target control of the inspired oxygen concentration (FIO2) and end-expired concentration (FA) of a potent inhaled anesthetic. İnitially before induction, we set the minimal fresh gas flow to 0.5 L min-1 and target end-expired agent concentration for 1 MAC (minimal alveolar concentration). Shortly after intubation of the patient, we switched to AGC mode.
  Interventions: Device: AGC mode
- Group Minimal Flow: İn this group; following intubation, we set the fresh gas flow to 4 L min-1 and than we readjusted fresh gas flow manually to 0.5 L min-1 after sevoflurane concentration reaching to 1 MAC.
- Group Medium Flow: İn this group; following intubation, we set the fresh gas flow to 4 L min-1 and than we readjusted fresh gas flow manually to 2 L min-1 after sevoflurane concentration reaching to 1 MAC.

INTERVENTIONS:
Device: AGC mode — Automated Gas Control mode at Maquet FLOW-i anesthesia machine
  Groups: Group AGC

SUMMARY:
The aim of this study was to compare the AGC mode and manually controlled minimal-flow anesthesia for volatile anesthetic consumption, hemodynamic parameters, and recovery from anesthesia

DETAILED DESCRIPTION:
Modern anesthesia machines use circular systems in which ventilated gas re-circulates to a certain degree and is therefore reused, preserving temperature, and humidity. The rebreathing fraction is increased by a reduction in fresh gas flow, which leads to a considerable decrease in consumption of fresh gas and volatile anesthetics, resulting in reductions in cost and atmospheric pollution. In a closed ventilation system, only the patient's requirements for oxygen and anesthetic agents are supplemented. A fresh gas flow-rate of 0.5 l/min is defined as the minimal-flow technique. The oxygen and anesthetic gas titration can be manually controlled by the anesthetist. To assure safe and appropriate anesthesia, manually controlled anesthesia requires constant monitoring and numerous adjustments to the gas dosage by the anesthetist, especially for low- and minimalflow anesthesia. Oxygen flow and volatile anesthetics can also be automatically controlled by anesthesia machines using end-tidal control (such as AGC mode of Maquet FLOW-i anesthesia machine), which ensures constant end-tidal concentration of oxygen and anesthetic gas via feedback and continuous automatic adjustment mechanisms. Anesthesiologists needing to make fewer interventions during a case may have clinical importance in terms of distraction, record keeping and patient safety. In addition to this advantage, we wanted to compare the AGC mode and manually controlled minimal-flow anesthesia for volatile anesthetic consumption, hemodynamic parameters, and recovery from anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* undergoing breast surgery
* ASA physical status I-II
* female
* operation lasting at least 1 hour
* those who agreed to volunteer for the study with an informed consent form

Exclusion Criteria:

* coronary artery disease, CHF
* pregnancy or breastfeeding women
* decompensated diabetes mellitus
* kidney or liver failure
* chronic obstructive pulmonary disease
* opioid sensitivity
* history of malignant hyperthermia
* history of smoking
* alcohol or drug addiction
* significant anemia
* sepsis
* BMI >35
* patients with allergies to the drugs used in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Between 18-65 years, female patients underwent breast surgery
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Consumption of Volatile Agent | during the surgery
  Difference of Sevoflurane Consumption between the groups

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Medicine Faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided